CLINICAL TRIAL: NCT04217902
Title: VOIES-D-ql (Visualization for the Optimization of Interactions and Experiences in Healthcare Services in Diabetes Care)
Brief Title: VOIES-D-ql - Qualitative Study on Experiences of Diabetes Care Delivery and Planning
Acronym: VOIES-D-ql
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0897
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Diabete Type 1; Diabete Type 2
Keywords: Diabete Type 1; Diabete Type 2; Diabete Care
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People living with diabetes in Grenoble and Lyon areas: Eligible patients with type 1 or type 2 diabetes 1) during or after hospitalization for decompensation, ketoacidosis, or other emergency or elective interventions such as insulin pump installation, 2) followed in routine care in specialized diabetes services, 3) participating in patient associations.
  Interventions: Other: Description of patients' experiences of diabetes care delivery and planning
- Health care professionals working in diabetes care in Grenoble: Health care professionals working with diabetes care in specialized services or ambulatory care.
  Interventions: Other: Description of health care professionals needs and experiences in diabetes care delivery and planning

INTERVENTIONS:
Other: Description of patients' experiences of diabetes care delivery and planning — Semi-directed interviews will be conducted with people living with type 1 or type 2 diabetes in person or by phone to assess and describe the care delivery pathway they have been through. Information on 3 domains will be assessed: clinical (information they consider essential for health care professionals to systematically have access to during consultations and other health-related interventions such as therapeutic education sessions), technological (what kind of digital services and technologies they use or are willing to use), and behavioural (the decision-making process and the key interactions that build the care delivery pathway).
  Groups: People living with diabetes in Grenoble and Lyon areas
Other: Description of health care professionals needs and experiences in diabetes care delivery and planning — Semi-directed interviews will be conducted with health care professionals working in diabetes care in person or by phone to assess and describe their needs and experiences in diabetes care. Information on 3 domains will be assessed: clinical (the information they consider to be essential to inform decisions in diabetes care, where and if they currently find that information and problems they might encounter), technological (which software they currently use and how data is input into clinical information systems), and behavioural (how care coordination is currently managed, how interactions with patients and other professionals are undertaken).
  Groups: Health care professionals working in diabetes care in Grenoble

SUMMARY:
Population aging and the increase in incidence and prevalence of potentially disabling chronic conditions make health care more and more complex and costly. In this context, timelines are longer and adherence to care provision and health status are more variable - both within and between patients - and care is provided by different health care professionals, as well as services outside the health system, which may work at various levels of service integration. For diabetes, this is especially the case: patients at high risk for multimorbidity interact with multiple health care professionals, such as primary care physicians, diabetes specialists, nurses, nutritionists and therapeutic educators, with different perspectives to treatment. The patient is frequently the only link between the different health care professionals, and very often the main source of information regarding performed procedures, diagnoses and treatment decisions.

A current challenge facing all health care stakeholders, including policy makers, practitioners, businesses, and patients, is to coordinate the available services and integrate care ensuring safety, effectiveness, and comprehensiveness in relation to the needs of individual users across the lifespan. Routine collected data can provide key information to completely assess a patient's health status and thus help evaluating and deciding adapted steps in treatment to stabilize or improve clinical outcomes.

In France, the Dossier Medical Partagé (Shared Medical Record) represents an effort to centralize and improve accessibility, to patients and professionals alike, of medical information. This system is yet little adopted and there is the need for added value initiatives to exploit the tool's potential. In other countries, like the UK, the governmental unit NHSX develops public policies and good practices for the digital transformation of the NHS. In the United States, working groups like the Health Information Technology Working Group, in the National Institute of Diabetes and Digestive and Kidney Diseases, develop electronic care plans using Electronic Health Record data for chronic kidney disease patients. These initiatives, among others, show the necessity of simple, visual communication in order to build a comprehensive care delivery pathway to inform decision and further care planning, according to health goals set by shared decision-making.

This study aims to describe individual experiences of chronic care delivery of people living with diabetes and also from healthcare professionals working in diabetes care from 3 different domains: clinical (relevant clinical criteria necessary for the decision-making process, goal setting and planning), technological (tools used in routine practice and in patients' daily lives), and behavioural (behaviours and interactions that build the patient's pathway and strategies implemented by patients and professionals to help the decision-making process).

Locations of the study : Primary and secondary healthcare facilities and patient associations in Lyon and Grenoble areas

ELIGIBILITY:
Inclusion Criteria:

Patient

* At least 18 years old
* Diagnosed with type 1 or type 2 diabetes according to HAS criteria and confirmed by and endocrinologist since at least one year
* Having had at least one consultation with a health care professional in the last 12 months
* Able to communicate in French
* Able to participate in an interview and not opposing to participate in the study

Professional

* Having at least one year of professional experience in diabetes care
* General practitioner, endocrinologist, diabetologist, intern, nurse, nutritionist or professional specialized in therapeutic education

Exclusion Criteria:

Patient

* Inability to communicate in French
* Institutionalized person

Professional

* Professional not having had at least one consultation with a person living with diabetes in the last 12 months

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People living with type 1 or type 2 diabetes recruited from Hospices Civils de Lyon or Centre Hospitalier Universitare Grenoble-Alpes, patient associations or online patient groups & HCPs
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Description of individual experiences of patients and health care professionals in diabetes care. | The moment of the interview (Day 0)
  Socioeconomic status will be assessed, health literacy using the Brief Health Literacy Screening (BHLS), and a semi-directed interview will be undertaken with people living with type 1 or type 2 diabetes. The latter aims t obtain a description of their experiences concerning how their care delivery pathways were built over time, how health-related decisions are made individually and what data they consider health care professionals they interact with should systematically have access to (considering the 3 domains previously described). Health care professionals will also be interviewed regarding their experiences and needs in diabetes care, in the shared decision-making process and in establishing care coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory HESPER EA 7425, University Claude Bernard Lyon 1, Lyon, France